CLINICAL TRIAL: NCT02254837
Title: Zilver PTX Post-Market Surveillance Study of Paclitaxel-Eluting Stents for Treating Femoropopliteal Artery Disease in Japan
Brief Title: Zilver PTX Post-Market Study in Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-005-PTX
Record Dates: First submitted 2014-09-24; First posted 2014-10-02 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zilver PTX (Experimental)
  Interventions: Device: Zilver PTX Drug-Eluting Stent

INTERVENTIONS:
Device: Zilver PTX Drug-Eluting Stent

SUMMARY:
Japanese post market clinical study of the Zilver PTX device.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic peripheral arterial disease (PAD) involving the above-the-knee femoropopliteal arteries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 909 (Actual)
Dates: Start 2012-05; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of stent fracture | 5 years
Rate of adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Dake, MD, Principal Investigator — Department of Cardiothoracic Surgery, Stanford University Medical Center, Stanford, CA

REFERENCES:
- [Derived] Sugimoto M, Komori K, Yokoi H, Ohki T, Kichikawa K, Nakamura M, Nanto S, O'Leary EE, Lottes AE, Saunders AT, Dake MD. Long-Term Effectiveness of a Drug-Eluting Stent for Femoropopliteal In-Stent Restenosis: Subanalysis of the Zilver PTX Japan Post-Market Surveillance Study. J Endovasc Ther. 2021 Apr;28(2):229-235. doi: 10.1177/1526602820966708. Epub 2020 Oct 21. PMID 33084502
- [Derived] Dake MD, Fanelli F, Lottes AE, O'Leary EE, Reichert H, Jiang X, Fu W, Iida O, Zen K, Schermerhorn M, Zeller T, Ansel GM. Prediction Model for Freedom from TLR from a Multi-study Analysis of Long-Term Results with the Zilver PTX Drug-Eluting Peripheral Stent. Cardiovasc Intervent Radiol. 2021 Feb;44(2):196-206. doi: 10.1007/s00270-020-02648-6. Epub 2020 Oct 6. PMID 33025243
- [Derived] Kichikawa K, Ichihashi S, Yokoi H, Ohki T, Nakamura M, Komori K, Nanto S, O'Leary EE, Lottes AE, Snyder SA, Dake MD. Zilver PTX Post-market Surveillance Study of Paclitaxel-Eluting Stents for Treating Femoropopliteal Artery Disease in Japan: 2-Year Results. Cardiovasc Intervent Radiol. 2019 Mar;42(3):358-364. doi: 10.1007/s00270-018-2110-1. Epub 2018 Nov 8. PMID 30411151
- [Derived] Yokoi H, Ohki T, Kichikawa K, Nakamura M, Komori K, Nanto S, O'Leary EE, Lottes AE, Snyder SA, Dake MD. Zilver PTX Post-Market Surveillance Study of Paclitaxel-Eluting Stents for Treating Femoropopliteal Artery Disease in Japan: 12-Month Results. JACC Cardiovasc Interv. 2016 Feb 8;9(3):271-277. doi: 10.1016/j.jcin.2015.09.035. PMID 26847118